CLINICAL TRIAL: NCT00423501
Title: A Double Blind, Placebo-controlled, Dose-ranging Study to Investigate the Effect on Glycemic Control, Safety, Pharmacokinetics and Pharmacodynamics of GLP-1 in Patients With Type 2 Diabetes Mellitus Treated With a Stable Dose of Metformin.
Brief Title: A Study of a GLP-1 Analogue in Patients With Type 2 Diabetes Treated With Metformin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20688
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: taspoglutide
- 2 (Experimental)
  Interventions: Drug: taspoglutide
- 3 (Experimental)
  Interventions: Drug: taspoglutide
- 4 (Experimental)
  Interventions: Drug: taspoglutide
- 5 (Experimental)
  Interventions: Drug: taspoglutide
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — sc weekly
  Arms: 6
Drug: taspoglutide — 20mg sc weekly
  Arms: 3
Drug: taspoglutide — 10mg sc every 2 weeks
  Arms: 4
Drug: taspoglutide — 5mg sc weekly
  Arms: 1
Drug: taspoglutide — 10mg sc weekly
  Arms: 2
Drug: taspoglutide — 20mg sc every 2 weeks
  Arms: 5

SUMMARY:
This 6 arm study will evaluate the efficacy, safety, pharmacokinetics and pharmacodynamics of multiple doses and regimens of a GLP-1 analogue in patients with type 2 diabetes who are treated with a stable dose of metformin. Patients will be randomized to receive either subcutaneous placebo, or subcutaneous GLP-1 analogue, 5mg, 10mg or 20mg weekly, or 10mg or 20mg every 2 weeks. All patients will continue on their existing metformin treatment regimen throughout the study. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes mellitus, with stable metformin treatment for >=3 months;
* stable weight +/-10% for >=3 months before screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* treatment with any anti-hyperglycemic medication other than metformin monotherapy during last 3 months;
* use of weight-lowering medications in the last 3 months;
* uncontrolled hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbAlc | Week 8

SECONDARY OUTCOMES:
Absolute change from baseline in FPG, fructosamine, body weight, fasting insulin, C-peptide, glucagon. | Week 8
Changes in lipid profile | Week 8
AEs, laboratory parameters, primary pharmacokinetic parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- United States (10):
  - Washington D.C., District of Columbia
  - Woodstock, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Rochester, New York
  - Portland, Oregon
  - Dallas, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Australia (2):
  - Adelaide
  - Camperdown
- Bulgaria (5):
  - Dimitrovgrad
  - Pleven
  - Rousse
  - Sofia
  - Varna
- Germany (7):
  - Bad Lauterberg im Harz
  - Berlin
  - Görlitz
  - Hanover
  - Mainz
  - Neuss
  - Nuremberg
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Mexico (4):
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
- Romania (8):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Jud Covasna
  - Mures
  - Ploieşti
  - Satu Mare
  - Sibiu

REFERENCES:
- [Derived] Nauck MA, Ratner RE, Kapitza C, Berria R, Boldrin M, Balena R. Treatment with the human once-weekly glucagon-like peptide-1 analog taspoglutide in combination with metformin improves glycemic control and lowers body weight in patients with type 2 diabetes inadequately controlled with metformin alone: a double-blind placebo-controlled study. Diabetes Care. 2009 Jul;32(7):1237-43. doi: 10.2337/dc08-1961. Epub 2009 Apr 14. PMID 19366970